CLINICAL TRIAL: NCT06249295
Title: The Efficacy of Postoperative Oral Cryotherapy in Sore Throat and Daily Life in Patients With Sleep Apnea
Brief Title: Postoperative Oral Cryotherapy in Sore Throat and Daily Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Hsiang Chu Pai, Principal Investigator, Chung Shan Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS1 21024
Record Dates: First submitted 2024-01-30; First posted 2024-02-08 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive sleep apnea syndrome; oral cryotherapy; pain; daily life
MeSH Terms: conditions — Sleep Apnea, Obstructive; Pain | interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: The experimental group used drinking water from a water dispenser with regular filter replacement and maintenance, plus a 2x5x7 cm (50 ml) ice lolly module to make ice lollies ,and then intervened in the post-surgical period using oral cold therapy (ice lolly in the mouth), while the control group received general routine care.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The experimental group used drinking water from a water dispenser with regular filter replacement and maintenance, plus a 2x5x7 cm (50 ml) ice lolly module to make ice lollies, and then intervened in the post-surgical period using oral cold therapy (ice lolly in the mouth).
  Interventions: Other: oral cryotherapy
- control group (No Intervention): The control group received general routine care.

INTERVENTIONS:
Other: oral cryotherapy — The experimental group used drinking water from a water dispenser with regular filter replacement and maintenance, plus a 2x5x7 cm (50 ml) ice lolly module to make ice lollies, and then intervened in the post-surgical period using oral cold therapy (ice lolly in the mouth)
  Arms: Intervention group

SUMMARY:
The purpose of this study will to evaluate the degree of postoperative sore throat and Life Impairment changes in patients with sleep apnea who underwent da Vinci robotic arm surgery as an intervention of oral cryotherapy.

DETAILED DESCRIPTION:
An experimental study was conducted with 32 patients in the experimental group and 32 patients in the control group. The experimental group used drinking water from a water dispenser with regular filter replacement and maintenance, plus a 2x5x7 cm (50 ml) ice lolly module to make ice lollies,and then intervened in the postsurgical period using oral cold therapy (ice lolly in the mouth),while the control group received general routine care. The control group received regular care. The assessment tools included the Pain Profile Scale and the Life Impairment Scale, and the assessment period was from the first day to the 14th day after the operation.

ELIGIBILITY:
Inclusion Criteria:

* (1)Admission age is 18 years or above, conscious, able to communicate in Mandarin and Taiwanese, and willing to be measured and fill out the questionnaire after explaining the process and purpose of the study.
* (2) The study was conducted in hospitalised patients diagnosed with sleep apnea who underwent surgery.

Exclusion Criteria:

* (1) Diagnostic diagnosis of the disease not clearly known.
* (2) Patients with unclear consciousness.
* (3) Patients who have been diagnosed with mental illness before the diagnosis of the -
* disease or recently diagnosed with mental illness.
* (4) People with paraplegia or low behavioural ability.
* (5) Patients who have suffered a stroke.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
sore throat | up to 2 weeks
  The Pain Profile Scale assesses the pain level of the patient, which consists of 8 items: total pain level, throat pain level, throat pain during swallowing, ear pain during swallowing, difficulty swallowing, limitation of physical activity, oral odor, and sleep disruption, and other symptoms related to pain. The scoring criteria are based on a four-point scale: 0 for no sensation, 1 for mild, 2 for The scale is based on a four-point scale: 0 for no sensation, 1 for mild, 2 for moderate, and 3 for severe to present a multidimensional pain assessment.

SECONDARY OUTCOMES:
daily life | up to 2 weeks
  The secondary outcome was to measure the extent to which the level of physical pain interfered with daily life, with a scale of 1 as not at all interfered, 2 as somewhat interfering, 3 as moderately interfering, 4 as considerably interfering, and 5 as extremely interfering, to understand the impact of pain on daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang Chu Pai, PhD, Study Director — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan